CLINICAL TRIAL: NCT05014893
Title: Neural Mechanisms of Cognitive Assessment and Rehabilitation for Cognitive Decline
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Center for Rehabilitation Technical Aids (Other)
Collaborators: Nanjing Brain Hospital (Unknown); The Third People's Hospital of Yunnan Province (Other Government); Central South University (Other); Beijing academy of science and technology (Unknown); Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Pengxu Wei, Director, National Research Center for Rehabilitation Technical Aids
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 201900045
Record Dates: First submitted 2021-08-01; First posted 2021-08-20 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Mild Cognitive Impairment (MCI); Subjective Cognitive Decline (SCD); Aging; Healthy
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control group, without specific treatments
- Cognitive training (Experimental): This group receives treatments to improve cognitive function.
  Interventions: Combination Product: multi-modal targeted intervention (e.g., cognitive training, exercise, games)

INTERVENTIONS:
Combination Product: multi-modal targeted intervention (e.g., cognitive training, exercise, games) — The Intervention group will be given recommended interventions tailored to individuals based on their risks (e.g., physical exercise programs, cognitive training, dietary advice, control of blood pressure and cholesterol, healthy diet, control obesity, stop smoking,reduce alcohol excess)
  Arms: Cognitive training

SUMMARY:
This study investigates the neural mechanisms of cognitive function decline, cognitive assessment methods for subjects with mild cognitive dysfunction (Mild cognitive impairment, MCI, or cognitive decline milder than MCI), and the approaches used to improve and restore cognitive function.

DETAILED DESCRIPTION:
Cognitive assessment tools are used to assess cognitive function of subjects in different cities. Functional and structural MRI and EEG are applied to investigate the neural mechanisms of cognitive function decline and effects of methods to improve and restore cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Adults being able to walk at least a block, and
* Adults with subjective cognitive decline (SCD), or
* Adults with mild cognitive impairment (MCI), or
* Adults with normal cognitive function

Exclusion Criteria:

* Clinical diagnosis of dementia
* Adults who cannot follow the protocal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Cognitive function (SCD-9) | Change from Baseline Cognitive test results at 3 months.
  The SCD-9 questionnaire is used to assess cognitive function of participants.
Change in Cognitive function (MoCA) | Change from Baseline Cognitive test results at 3 months.
  The Montreal Cognitive Assessment test is used to assess cognitive function of participants.
Change in Cognitive function (AD8) | Change from Baseline Cognitive test results at 3 months.
  The AD8 test is used to assess cognitive function of participants.
Change in Cognitive function (CDR) | Change from Baseline Cognitive test results at 3 months.
  The Clinical Dementia Rating (CDR) test is used to assess cognitive function of participants.

SECONDARY OUTCOMES:
Change in Physical capacity (TUG) | Change from Baseline physical capacity test results at 3 months.
  The timed up and go (TUG) test is used to evaluate physical capacity of participants.
Change in Physical capacity (chair standing) | Change from Baseline physical capacity test results at 3 months.
  The 30-second chair standing test is used to evaluate physical capacity of participants.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 24 months.
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Pengxu Wei, Principal Investigator — National Research Center for Rehabilitation Technical Aids
Locations (1):
- National Research Center for Rehabilitation Technical Aids, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No